CLINICAL TRIAL: NCT01065961
Title: Prospective Randomized Controlled Trail of the Effects of Steroids on Swallowing, Airway and Arthrodesis Related to Myulti-Level Anterior Cervical Reconstruction
Brief Title: Randomized Controlled Trials of the Effects of Decadron on Swallowing, Airway, and Arthrodesis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Darryl DiRisio, MD, Albany Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D-01
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2008-11

CONDITIONS: Swallowing
Keywords: anterior; cervical; fusion; swallowing; Swallowing after anterior cervical discectomy and fusion; Bony fusion rates post anterior cervical discectomy and fusion
MeSH Terms: interventions — Calcium Dobesilate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decadron (Active Comparator): Subject will be given Decadron 0.2mg/kg intraoperatively. This dose will be followed by 4 mg. every 6 hours for the first 24 hours.
  Interventions: Drug: Decadron
- Saline (Placebo Comparator): subject will be given a blinded dose of placebo saline intraoperatively followed by placebo doses every 6 hours for 24 hours.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Decadron — Decadron will be given at a dose of 0.2 mg/kg intraoperatively, followed by Decadron 4 mg. every 6 hours for 24 hours.
  Arms: Decadron
Drug: Saline — Placebo saline will be given intraoperatively as well as 4 doses every 6 hours for 24 hours.
  Arms: Saline

SUMMARY:
Anterior cervical discectomy and fusion with or without decompression is a well-established surgical treatment for spine patients with the appropriate indications. Anterior approach involves some retraction that affect the midline structures of the anterior neck. Irritation and swelling may result, leading to postoperative dysphagia and the less common but critically important occurrence of postoperative airway compromise. Steroids given intraoperatively may reduce the incidence of these adverse outcomes by reducing the degree of swelling within the anterior neck subsequent to local surgical tissue trauma.

The investigators hypothesize that the use of steroids intraoperatively provides a significant benefit to the patient, in terms of reduced incidence of dysphagia and airway compromise.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Cervical spondylosis requiring surgical treatment at 2 or more motion segments
* Ventrally - approachable vertebral levels

Exclusion Criteria:

* Minors (under 18 years old)
* Pregnant women
* Patients currently taking steroids
* Patients requiring surgical treatment at only one segment
* Comatose or incapacitated patients who cannot consent to participate
* Wards of the state
* Persons with an allergy to dexamethasone or related drugs
* Persons employed at Albany Medical Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
subjects will demonstrate good bony fusion | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center, Albany, New York, United States

REFERENCES:
- [Derived] Jeyamohan SB, Kenning TJ, Petronis KA, Feustel PJ, Drazin D, DiRisio DJ. Effect of steroid use in anterior cervical discectomy and fusion: a randomized controlled trial. J Neurosurg Spine. 2015 Aug;23(2):137-43. doi: 10.3171/2014.12.SPINE14477. Epub 2015 May 1. PMID 25932600